CLINICAL TRIAL: NCT07112703
Title: Effect of Incentive Respiratory Training on Pulmonary Functions and Functional Capacity in Children With B-thalassemia Major
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rawan Mohammed Khairy Mostafa Elsawy (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Rawan Mohammed Khairy Mostafa Elsawy, rawan mohamed khairy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rawan_Phd
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Incentive Spirometer; Pulmonary Function; Functional Capacity; Child, Only; Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditional breathing exercise (Active Comparator): 20 children will receive traditional breathing exercise for 30 minutes 2 times per month for 3 months.
  Interventions: Other: Diaphragmatic breathing; Other: Pursed lip breathing:; Other: Costal breathing exercises
- traditional breathing exercise and incentive spirometer breathing (Experimental): 20 children who will receive traditional breathing exercise for 15 minutes and breathing exercises by incentive spirometer for 15 minutes 2 times per month for 3 months
  Interventions: Other: Incentive spirometer exercises; Other: Diaphragmatic breathing; Other: Pursed lip breathing:; Other: Costal breathing exercises

INTERVENTIONS:
Other: Incentive spirometer exercises — The study group was instructed to use an incentive spirometer, which should be held upright, sealed around the mouthpiece, and taken slowly and deep breaths. They will be motivated to achieve a preset volume through visual feedback. The child will hold their breath for 2-3 seconds at full inspiration and, after each set of 10 breaths, cough to clear mucus from the lungs. The exercise duration is 15 minutes.
  Arms: traditional breathing exercise and incentive spirometer breathing
Other: Diaphragmatic breathing — The child will lie on their back, place one hand on their belly and one on their chest, and use a balloon or doll to fill both belly and chest up like a balloon. Inhale deeply, let the hands on the belly rise, then exhale slowly, making the belly down. The exercise will last for 10 minutes.
Other: Pursed lip breathing: — Sit in a seated position with crossed legs or knees. Inhale slowly through the nose for three seconds, then exhale through pursed lips, similar to blowing out birthday candles.
Other: Costal breathing exercises — The study involves conducting Costal breathing exercises for children. The exercises involve placing hands on the apical region of the lung, turning the child's head, relaxing the shoulder and neck muscles, taking a deep breath, pushing the hand out, holding, and exhaling slowly. The hands provide pressure and resistance after initiation of inspiration, and the children rest for 2 minutes between exercises. The duration of the exercise varies between the control and study groups.

SUMMARY:
The study was done to:

1. Investigate the effect of respiratory training on functional lung capacity and
2. To detect the effect of respiratory training on pulmonary functions in children with β-thalassemia major.
3. To detect the level of oxygen saturation and heart rate during and after blood transfusion in children with β-thalassemia major.

DETAILED DESCRIPTION:
Children with thalassemia require regular blood transfusions, which can lead to complications and affect lung capacity, oxygen saturation, and heart rate. To improve lung function capacity, this study aims to enhance physical fitness for children with B-thalassemia major, enabling optimal performance in daily activities and leisure activities. Physical activity focused on fitness is essential for children to find pleasure in physical activities and improve oxygen saturation levels. This study may also help physiotherapists understand the importance of improving lung function capacity for children with B-major thalassemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as thalassemia & subjected to blood transfusion
2. Their age range from 6 to 10 years old
3. Both sexes, male and female, will participate.
4. Subjects are able to follow simple verbal commands or instructions included in the procedures.

Exclusion Criteria:

1. Children with mental retardation or any other disability .
2. Children with visual or hearing defects.
3. Children with cardiovascular, chest pulmonary, and heart diseases.
4. Children with any postoperative cardiovascular, chest pulmonary, and heart conditions.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
assessment of oxygen saturation | before exercises and immediately after blood transfusion
  A child should rest for five minutes before taking an oximeter reading. The meter should be placed on the child's fingertip, and if the numbers fluctuate, the oxygen saturation level will be clearly labeled on the screen device.
assessment of heart rate | before exercises and immediately after blood transfusion
  A child should rest for five minutes before taking an oximeter reading. The meter should be placed on the child's fingertip, and if the numbers fluctuate, the heart rate level will be clearly labeled on the screen device.

SECONDARY OUTCOMES:
assessment of slow vital capacity | before exercises and immediately after blood transfusion
  Using neuro-soft spirometer. The process involves calibrating an instrument, data entry, and child preparation for measurements. Calibration involves removing the mouthpiece, attaching it to the flow sensor, and adjusting the device pump. Data entry involves sterilizing the mouthpiece and entering patient information. Assessment procedures involve sitting comfortably, recording data, performing test maneuvers, and repeating the test if results aren't acceptable.
  The child is instructed to take two to three normal breaths, exhale slowly and inhale gently, with a diagram displayed on the screen to measure their breathing strength. The record icon is closed after the test, and 1-2 minutes of rest is allowed between measurements.
assessment of forced expiration | before exercises and immediately after blood transfusion
  Using neuro-soft spirometer. The process involves calibrating an instrument, data entry, and child preparation for measurements. Calibration involves removing the mouthpiece, attaching it to the flow sensor, and adjusting the device pump. Data entry involves sterilizing the mouthpiece and entering patient information. Assessment procedures involve sitting comfortably, recording data, performing test maneuvers, and repeating the test if results aren't acceptable.
  A forced expiration test involves a child taking two to three breaths, inhaling deeply, and blowing air through the mouthpiece until no air is left. A candle is shown on the screen to motivate the child. The test is repeated three times, and the record icon is closed.
assessment of Maximal voluntary ventilation test | before exercises and immediately after blood transfusion
  Using neuro-soft spirometer. The process involves calibrating an instrument, data entry, and child preparation for measurements. Calibration involves removing the mouthpiece, attaching it to the flow sensor, and adjusting the device pump. Data entry involves sterilizing the mouthpiece and entering patient information. Assessment procedures involve sitting comfortably, recording data, performing test maneuvers, and repeating the test if results aren't acceptable.
  A maximal voluntary ventilation test is conducted by inhaling and exhaling rapidly for 10 seconds, with a diagram showing inspiration and expiration strength. The record icon is closed after 10 seconds, and the test is repeated three times.
Assessment of functional capacity: | before exercises and immediately after blood transfusion
  The study uses a six-minute walk test to assess children's functional capacity. The child walks on a 10 meter unobstructed path, with a therapist monitoring their progress. They cover as many turns as possible without running. Chairs are placed at each 5 meter distance for rest and recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university hospitals., Zagazig, Egypt